CLINICAL TRIAL: NCT03152799
Title: Remote Ischaemic Conditioning in Endovascular Recanalization for Proximal Anterior Circulation Occlusion (RICE PAC) Study
Brief Title: Remote Ischaemic Conditioning in Endovascular Recanalization for Proximal Anterior Circulation Occlusion Study
Acronym: RICE PAC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other); National Hospital for Neurology and Neurosurgery (NHNN) at Queen Square (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 222254
Record Dates: First submitted 2017-03-08; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Ischemic Stroke
Keywords: remote ischaemic conditioning; remote ischemic conditioning; cerebral infarction; ischaemia reperfusion injury; ischemia reperfusion injury; anterior circulation stroke; mechanical thrombectomy
MeSH Terms: conditions — Ischemic Stroke; Cerebral Infarction; Reperfusion Injury

STUDY DESIGN:
Intervention Model Description: pilot, single-centre, double-blind, sham-controlled (non-clinical trial of investigational medicinal product [non-CTIMP]) study of repeated daily remote ischaemic conditioning vs placebo/sham in the context of acute anterior circulation stroke
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, Care Provider / Clinician Health Professional, Investigator, and Outcomes assessors will be blinded to the allocation and randomisation of study participatants. It is anticipated that
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischaemic Pre-Conditioning (RIPC) Intervention (Experimental): Remote Ischaemic Pre-Conditioning intervention to be applied via peripheral blood pressure cuff inflation/deflations to upper lower limb contra-lateral to affected side of hemiparesis
  Interventions: Procedure: RIPC Remote Ischaemic Pre-Conditioning
- Sham Control (Sham Comparator): Sham Control to be applied via peripheral blood pressure cuff inflation/deflations to upper lower limb contra-lateral to affected side of hemiparesis
  Interventions: Other: Sham Control

INTERVENTIONS:
Procedure: RIPC Remote Ischaemic Pre-Conditioning — intermittent limb ischaemia via a peripheral blood pressure cuff inflation and deflation
  Other Names: Remote Ischaemic PreConditioning
  Arms: Remote Ischaemic Pre-Conditioning (RIPC) Intervention
Other: Sham Control — intermittent peripheral blood pressure cuff inflation and deflation which does not induce a protective cellular response
  Arms: Sham Control

SUMMARY:
Ischaemic stroke causes significant morbidity and mortality and is a leading cause of disability within an ageing United Kingdom (UK) population. Proximal anterior circulation occlusion is associated with a particularly poor prognosis, but its management has undergone a paradigm shift following clinical introduction of endovascular recanalization, establishing rapid reperfusion of the ischaemic penumbra.

Remote ischaemic conditioning (RIC) is highly effective at attenuating cerebral infarction in basic research studies and has the potential to further improve patient outcome if used as an adjunct to invasive revascularisation strategies. We aim to trial remote ischaemic conditioning at the time of revascularisation, and then daily for the duration of the seven-day in-patient stay, compared to a sham conditioning procedure. This pilot, single-centre study will determine efficacy/ tolerability of RIC to reduce cerebral infarction (primary endpoint: determined by brain magnetic resonance imaging [MRI]) and improve functional status (secondary end-points: National Institutes of Health Stroke Severity (NIHSS); European Quality of Life questionnaire EurQoL), with the data providing the necessary parameters for power calculations and leveraging charitable funding for a subsequent multi-centre study.

DETAILED DESCRIPTION:
The aims of our study are to:

1. Demonstrate safety of remote ischaemic conditioning (RIC) in stroke patients;
2. Demonstrate practicality of the intervention (RIC);
3. Demonstrate the practicality of the study protocol and imaging modalities;
4. Determining appropriate and measurable end-points: e.g. cerebral infarct reduction (MRI), reduction of cerebral oedema, functional assessment and quality of life survey;
5. Provide preliminary data on likely effect size of the RIC intervention versus the sham procedure.

Background and Rationale:

Acute ischaemic stroke represents a significant cause of morbidity and mortality in the UK. It is estimated that 110,000 strokes occur in England each year, with an incidence of between 1-36/1000/year. Patients presenting with a proximal vessel occlusion in the anterior circulation have a particularly poor prognosis, with approximately 20% 90-day mortality and significant morbidity despite thrombolysis. Recently, endovascular recanalization with mechanical thrombectomy trials have brought about a paradigm shift in the optimal management of this high-risk group of patients; the interventional extraction of the occluding thrombus demonstrating significant benefits in MR-CLEAN(3), ESCAPE, EXTEND-IA (intra-arterial), SWIFT PRIME and REVASCAT (revascularisation) studies. Echoing primary percutaneous intervention in the management of ST-elevation myocardial infarction, endovascular recanalization represents rapid restoration of blood flow to the ischaemic cerebrum - with the promise of improved neurological salvage and functional outcome.

Reperfusion Injury:

Reperfusion is not, however, a benign process. Demonstrable in many organ systems including the brain (but studied most extensively in the heart), reperfusion leads to rapid restoration of intracellular pH, mitochondrial calcium overload and generation of reactive oxygen species - conditions that are prime for the opening of the mitochondrial permeability transition pore (mPTP). The mPTP, a large capacitance pore that forms on the inner mitochondrial membrane, leads to mitochondrial disruption and the release of proteins that trigger cell death. Therefore modifying conditions of reperfusion/ triggering cellular protection pathways are the key targets for optimising tissue salvage associated with reperfusion following any acute revascularisation intervention.

Remote ischaemic conditioning:

The brain has been demonstrated to share many of the cytoprotective signalling pathways found in other organs such as the heart, and like the heart, can be protected by ischaemic conditioning(6). Ischaemic conditioning can be either applied either directly to the organ, or more conveniently to a remote tissue (such as an arm, through inflation of a blood pressure cuff), either prior to, during or immediately following the restoration of blood flow to the ischaemic tissue (pre-, peri- and post-conditioning respectively). The remote conditioning stimulus leads to the activation of cellular survival kinases (termed the reperfusion injury salvage kinase (RISK) cascade) that in turn leads to inhibition of mPTP opening, and thus cell survival.

Ischaemic conditioning and neuro-protection:

While the phenomenon of ischaemic conditioning was first described and best characterised in the heart, it is well recognised that the ischaemic conditioning can result in cytoprotection across many mammalian organs, including the brain. Indeed, contemporaneous with the seminal myocardial preconditioning paper by Reimer, Murray and Jennings in the dog, Schurr et al demonstrated ischaemic preconditioning could also protect adult rat hippocampal slices against injurious anoxia/re-oxygenation. Ischaemic conditioning of neuronal tissue has subsequently been demonstrated to be triggered and mediated by similar receptor and downstream signalling pathways (e.g. G-protein coupled receptors, RISK pathway activation and suppression of cell death pathways), and that remote ischaemic conditioning is also effective at significantly attenuating the volume of cerebral necrosis in rat experimental models of acute right middle cerebral artery occlusion stroke (typically reducing infarct size by 40-60%). Similar results are observed in mouse (middle cerebral embolization, followed by thrombolysis with tissue-plasminogen activator) and in piglet, where the injurious effects of hypothermic circulatory arrest were attenuated, improving both functional and histological outcomes.

With building evidence of efficacy against cerebral ischaemia/reperfusion injury in the pre-clinical basic science studies, there is enthusiasm to translate these encouraging data into an effective clinical strategy for the management of acute stroke in man. A recent prospective, open-label, blinded outcome proof-of-concept study in Danish patients undertook ischaemic per-conditioning in patients presenting with an acute stroke syndrome. With the conditioning stimulus performed in the ambulance, the ischaemic stroke diagnosis was made/confirmed later in hospital. In patients with confirmed ischaemic stroke, they found patients in the intervention arm had a better functional status by National Institutes of Health Stroke Scale score on admission and an overall smaller infarct, but the study was overall neutral on the pre-specified primary endpoint (penumbral salvage, defined as the volume of the perfusion-diffusion mismatch not progressing to infarction after 1 month). There are useful lessons and observations to be made regarding the design of this trial that influences the design of the trial proposed within this application. First, thrombolysis does not guarantee re-canalisation of the culprit artery, and where restoration of blood flow does occur, the time of onset of reperfusion may be unpredictable. Thus, restoration of blood flow may either not have occurred, or when it had, may have occurred outside the protective time-frame of the remote ischaemic conditioning stimulus (classical conditioning has a protective "window" of typically just 2-3 hours).

Therefore, we are seeking to combine ischaemic conditioning with an effective endovascular re-canalisation procedure where the success and time of reperfusion are known. Second, in the Danish study, there would have been significant heterogeneity in aetiology of the presenting stroke symptoms that will include both anterior and posterior circulation occlusion and also small vessel disease. The pre-clinical efficacy of remote ischaemic conditioning is predominantly with models of anterior circulation occlusion and therefore, we have made this cohort of patients the focus of our study. And finally, there is emerging evidence that in order to ensure persistent infarct size reduction, it is critical to combine both initial ischaemic per-conditioning and subsequent post-conditioning to tackle both the acute reperfusion injury (the first 15 minutes of reperfusion) and the subsequent second phase of reperfusion injury (that occurs in the following hours and days). Thus our study is designed to combine both ischaemic per-conditioning and repeated post-conditioning over the following seven days to harvest the benefit of both conditioning strategies.

Interestingly, a Chinese study (RIC to both arms daily for 300 days after the initial stroke) was shown to be safe and effective. While this study had a different outcome to ours (attenuating the rate of stroke recurrence following the initial presentation), the efficacy of the RIC intervention nonetheless provides further encouragement that RIC may be an effective intervention in this group of patients.

In summary therefore, we are seeking to combine ischaemic conditioning with an effective endovascular re-canalisation procedure where the success and time of reperfusion are known, in a vascular territory that is known to benefit from RIC and are looking to combine both ischaemic per-conditioning and repeated post-conditioning over the following seven days to harvest the benefit of both conditioning strategies upon acute and inflammatory phases of reperfusion injury - encompassing the period over which peak cerebral oedema is typically observed.

ELIGIBILITY:
Inclusion Criteria:

* Acute, symptomatic proximal anterior circulation occlusion
* able to commence remote ischaemic conditioning within 6h of symptom onset
* identified as candidate for endovascular intervention according to local criteria

Exclusion Criteria:

* Age < 18 years
* Coagulopathy; International Normalised Ratio (INR) >2, alteplase dose > 90mg or 0.9mg/kg; platelet count < 50 x 10^9/L
* pregnancy
* BP >= 185/110 despite therapeutic intervention
* medical illness which interferes with outcome assessments (disability from other neurological disease)
* dependent on others for activities of daily living (ADLs) prior to current stroke (mRS modified Rankin Score was 3 - 5).
* unlikely to be able to participate in study follow-up procedures (lives > 100 miles away; no fixed abode)
* already enrolled in another clinical trial involving investigational medicinal product or device
* baseline scan demonstrating significant prior infarction in the affected Middle Cerebral Artery (MCA) territory or an infarct that exceeds > 1/3 MCA territory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
reduction of infarct size as proportion of ischaemic penumbra following revascularisation | 3 months after revascularisation / thrombectomy
  Proportion of ischaemic penumbra determined by MRI at 3 months post-revascularisation

SECONDARY OUTCOMES:
Reduction of cerebral oedema and infarct size (second-phase reperfusion injury) | MRI at 7 days post-thrombectomy
  Proportion of ischaemic penumbra comparing MRI data at 24 hours and 7 days post-thrombectomy
Neurological Recovery at 24 h and 3 months post-revascularisation | at 24h hours and 3 months post-revascularisation
  modified Rankin Score
Neurological Recovery at 24 h and 3 months post-revascularisation | at 24h hours and 3 months post-revascularisation
  NIHSS (National Institutes of Health Stroke Scale)
Neurological Recovery at 24 h and 3 months post-revascularisation | at 24h hours and 3 months post-revascularisation
  QoL (Quality of Life) assessment

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Bell, PhD MRCP, Principal Investigator — Hatter Cardiovascular Institute UCL; Derek Yellon, PhD DSc, Study Director — Hatter Cardiovascular Institute UCL

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Department of Health: Progress in Improving Stroke Care. In: Office NA, editor.: The Stationary Office; 2010.
- [Background] Hippisley-Cox J, Pringle M, Ryan R. Stroke: Prevalence, Incidence and Care in General Practices 2002-2004. Final Report to the National Stroke Audit Team. In: Physicians RCo, editor. 2004.
- [Background] Berkhemer OA, Fransen PS, Beumer D, van den Berg LA, Lingsma HF, Yoo AJ, Schonewille WJ, Vos JA, Nederkoorn PJ, Wermer MJ, van Walderveen MA, Staals J, Hofmeijer J, van Oostayen JA, Lycklama a Nijeholt GJ, Boiten J, Brouwer PA, Emmer BJ, de Bruijn SF, van Dijk LC, Kappelle LJ, Lo RH, van Dijk EJ, de Vries J, de Kort PL, van Rooij WJ, van den Berg JS, van Hasselt BA, Aerden LA, Dallinga RJ, Visser MC, Bot JC, Vroomen PC, Eshghi O, Schreuder TH, Heijboer RJ, Keizer K, Tielbeek AV, den Hertog HM, Gerrits DG, van den Berg-Vos RM, Karas GB, Steyerberg EW, Flach HZ, Marquering HA, Sprengers ME, Jenniskens SF, Beenen LF, van den Berg R, Koudstaal PJ, van Zwam WH, Roos YB, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW; MR CLEAN Investigators. A randomized trial of intraarterial treatment for acute ischemic stroke. N Engl J Med. 2015 Jan 1;372(1):11-20. doi: 10.1056/NEJMoa1411587. Epub 2014 Dec 17. PMID 25517348
- [Background] Moore JM, Griessenauer CJ, Gupta R, Adeeb N, Patel AS, Ogilvy CS, Thomas AJ. Landmark papers in cerebrovascular neurosurgery 2015. Clin Neurol Neurosurg. 2016 Sep;148:22-8. doi: 10.1016/j.clineuro.2016.06.007. Epub 2016 Jun 18. PMID 27366977
- [Background] Bell RM, Yellon DM. There is more to life than revascularization: therapeutic targeting of myocardial ischemia/reperfusion injury. Cardiovasc Ther. 2011 Dec;29(6):e67-79. doi: 10.1111/j.1755-5922.2010.00190.x. Epub 2010 Jul 14. PMID 20645988
- [Background] Hahn CD, Manlhiot C, Schmidt MR, Nielsen TT, Redington AN. Remote ischemic per-conditioning: a novel therapy for acute stroke? Stroke. 2011 Oct;42(10):2960-2. doi: 10.1161/STROKEAHA.111.622340. Epub 2011 Aug 11. PMID 21836089
- [Background] Hougaard KD, Hjort N, Zeidler D, Sorensen L, Norgaard A, Hansen TM, von Weitzel-Mudersbach P, Simonsen CZ, Damgaard D, Gottrup H, Svendsen K, Rasmussen PV, Ribe LR, Mikkelsen IK, Nagenthiraja K, Cho TH, Redington AN, Botker HE, Ostergaard L, Mouridsen K, Andersen G. Remote ischemic perconditioning as an adjunct therapy to thrombolysis in patients with acute ischemic stroke: a randomized trial. Stroke. 2014 Jan;45(1):159-67. doi: 10.1161/STROKEAHA.113.001346. Epub 2013 Nov 7. PMID 24203849
- [Background] Ren C, Wang P, Wang B, Li N, Li W, Zhang C, Jin K, Ji X. Limb remote ischemic per-conditioning in combination with post-conditioning reduces brain damage and promotes neuroglobin expression in the rat brain after ischemic stroke. Restor Neurol Neurosci. 2015;33(3):369-79. doi: 10.3233/RNN-140413. PMID 25868435
- [Background] Meng R, Asmaro K, Meng L, Liu Y, Ma C, Xi C, Li G, Ren C, Luo Y, Ling F, Jia J, Hua Y, Wang X, Ding Y, Lo EH, Ji X. Upper limb ischemic preconditioning prevents recurrent stroke in intracranial arterial stenosis. Neurology. 2012 Oct 30;79(18):1853-61. doi: 10.1212/WNL.0b013e318271f76a. Epub 2012 Oct 3. PMID 23035060
- See also: Hatter Cardiovascular Institute — http://www.ucl.ac.uk/hatter-cardiovascular-institute/